CLINICAL TRIAL: NCT00595959
Title: CLiRpath® Excimer Laser System to Enlarge Lumen Openings
Brief Title: CELLO - CLiRpath® Excimer Laser System to Enlarge Lumen Openings
Acronym: CELLO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Rajesh M. Dave, M.D., Pinnacle Health Hospital, Central Pennsylvania Research Foundation
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9000-0001-03 CELLO
Record Dates: First submitted 2008-01-04; First posted 2008-01-16 (Estimated); Results first posted 2009-06-19 (Estimated); Last update posted 2011-07-12 (Estimated); Status verified 2011-06

CONDITIONS: Peripheral Artery Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Laser Treatment (Experimental): CLiRpath Photoablation Atherectomy System
  Interventions: Device: CLiRpath Photoablation System

INTERVENTIONS:
Device: CLiRpath Photoablation System — Use of CLiRpath Laser Catheter to improve vessel lumen diameter.

SUMMARY:
The objective of this study is to evaluate the safety and efficacy of the CLiRpath® Photoablation Atherectomy System consisting of the Bias Sheath guiding catheter, in combination with the available CLiRpath® Excimer Laser Catheters ≤ 2.0 mm, to create larger lumens for treatment within the superficial femoral and popliteal arteries above the knee.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Peripheral vascular disease Rutherford Classification 1, 2, or 3;
2. Eligible for revascularization of native vessel (PTA or bypass);
3. Willing and able to comply with the specified evaluations during hospitalization and all required follow-up examinations;
4. Written informed consent given before execution of study procedures; and
5. Age > 18 and ≤ 85 years.

Angiographic Inclusion Criteria

1. Reference vessel diameter >/= 4.0 mm and ≤ 7.0 mm as determined by physician visual angiographic assessment of the most normally appearing vessel segment within 10 mm proximal AND 10 mm distal to the target segment.
2. Stenosis within the SFA and/or popliteal artery above the knee of >/= 70% and </= 100% DS (occlusion), as determined by visual angiographic assessment by the investigator at the time of the procedure and documented by angiography in at least two (2) orthogonal views.
3. At least 1.0 cm of visible SFA stump beyond the origin of the profunda artery.
4. Total lesion length >/= 1.0 cm and ≤ 15.0 cm as determined by visual angiographic assessment at the time of the procedure, separate multiple lesions can be combined as two separate treatment areas as long as the sum total of all lesion lengths and/or treatment areas does not exceed 1.0 cm to 15.0 cm.
5. Patency (< 50% DS) of at least one (1) infrapopliteal artery in continuity with the native femoropopliteal artery.

   -

Exclusion Criteria:

General Exclusion Criteria

1. Contraindication to intravenous contrast material, heparin, aspirin or other medications required for a percutaneous interventional procedure;
2. Known bleeding or hyper-coagulation disorder;
3. Serum creatinine > 2.0 mg/dL;
4. Uncompensated congestive heart failure;
5. Current enrollment in any investigational study wherein patient participation has not been completed;
6. Prior enrollment in this study;
7. Suspected or confirmed pregnancy;
8. Any patient, who in the opinion of the investigator, would not be a good candidate for enrollment;
9. Myocardial infarction within 60 days; and
10. CVA/TIA within 60 days. Angiographic Exclusion Criteria

1.

1. Subintimal guidewire placement following pilot channel creation through a stenosis or occlusion with any excimer laser catheter, as visualized with IVUS;
2. Calcification likely to prevent the passage of the excimer laser catheter or CLiRpath® Photoablation Atherectomy system;
3. Ipsilateral and/or contralateral iliac stenosis >/= 50% DS that is not treated prior to enrollment in this study;
4. Ipsilateral and/or contralateral iliac treatment of a stenosis prior to enrollment with final residual stenosis >/= 30%, as determined in at least two (2) orthogonal views and documented by angiography;
5. Iliac treatment prior to enrollment where a perforation occurred requiring a covered stent, blood transfusion, or surgery for treatment of the perforation;
6. Identification of any lesion above the knee and/or below the knee in the treated leg (ipsilateral) that will require preplanned or predicted treatment within six (6) months after enrollment and prior to the completion of the six (6) month follow-up, including the iliac artery, the common femoral artery, the peroneal, anterior tibial, or posterior tibial arteries, or any area from the iliacs to the foot outside of the treatment area;
7. Lesions proximal and distal to the treatment site that are >/= 50% DS at time of enrollment;
8. Contralateral leg disease that requires treatment within the next 30 days and prior to completion of the 30 day follow-up;
9. Cardiovascular surgical or cardiovascular interventional procedures (including, but not limited to, aortic, renal, cardiac, carotid, femoro-popliteal, and below the knee) within 30 days prior to enrollment in this study;
10. Planned or predicted cardiovascular surgical or interventional procedures outside of the ipsilateral leg (including, but not limited to aortic, renal, cardiac, carotid, contralateral femoro-popliteal, and contralateral below the knee) within 30 days after entry into this study, and prior to completion of the 30-day follow-up; and
11. Perforation or dissection of grade "C" or greater seen during or after the creation of the pilot channel.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2006-11; Primary Completion 2007-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas M Rasmussen, Study Director — Spectranetics Corp.; Rajesh Dave, MD, Principal Investigator — Pinnacle Health Hospital, Central Pennsylvania Research Foundation

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from investigator patient referral base. Recruitment occurred between November 2006 and March 2007
Pre-assignment Details: Patients were screened for inclusion/exclusion criteria
Period: Overall Study
Arm/Group | Laser Treatment
Started | 65
Completed | 63
Not Completed | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
Age Continuous [Mean (Standard Deviation); unit: years] | 68.3 (10.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 39
Region of Enrollment [Number; unit: participants]
  United States | 65
Race/Ethnicity [Number; unit: participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 49
  African American | 11

OUTCOME MEASURES:

1. Primary Outcome: Laser Success
Description: The primary efficacy endpoint is laser success, defined as achieving >/= 20% average reduction in the percent (%) diameter stenosis, post-laser and prior to adjunctive therapy, based on angiographic core laboratory assessment.
Time Frame: Measured at time of procedure
Population: Per protocol
Measure: Mean (Standard Deviation); unit: percent reduction
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
percent reduction | 34.7 (17.8)
Statistical Analysis 1: Comparison: Laser Treatment; Comparing to an expected value of 20% reduction from initial to post-laser; Test type: Superiority or Other; p = 0.001, t-test, 1 sided — No adjustments

2. Primary Outcome: Major Adverse Events
Description: The primary safety endpoint is the occurrence of major adverse events defined as clinical perforation, major dissection requiring surgery, major amputation, cerebrovascular accidents (CVA), myocardial infarction, and death.
Time Frame: From discharge through the 6 month follow-up
Measure: Number; unit: events
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
events | 0

3. Secondary Outcome: Procedural Success
Description: Acute procedural success, defined as achievement of </= 30% final residual stenosis, as visually assessed by angiography after all adjunctive treatment(s) deemed necessary by the treating physician. Measures % of patients who achieved a final residual stenosis of </=30%.
Time Frame: measured at time of procedure
Population: Per protocol. All enrolled patients
Measure: Number; unit: percent with </=30% RS
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
percent with </=30% RS | 98.5

4. Secondary Outcome: Minimum and Maximum Lumen Diameters
Description: Minimum and maximum lumen diameters immediately after treatment with the CLiRpath® Photoablation Atherectomy System as determined by Intravascular Ultrasound (IVUS).
Time Frame: measured at time of procedure
Population: Analysis per protocol
Measure: Mean (Standard Deviation); unit: millimeters
Arm/Group | Laser Treatment
Number analyzed (Participants) | 48
millimeters
  Post pilot channel max lumen diameter | 4.2 (1.1)
  Post Turbo-Booster max lumen diameter | 5.1 (0.8)
  Post pilot channel min lumen diameter | 1.9 (0.6)
  Post Turbo-Booster min lumen diameter | 2.2 (0.8)

5. Secondary Outcome: Clinical Success
Description: Clinical success, defined as primary patency (≤ 50% stenosis at the treatment site), as assessed by duplex Doppler ultrasound at 30 days, six (6) months and 12 months post-procedure
Time Frame: measured post discharge thorugh 12 Months follow-up
Population: 65 patients at 30 days; 59 at 6 months; 46 at 12 months
Measure: Number; unit: percent of patients
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
percent of patients
  30 days; n=65 | 96.9
  6 months; n=59 | 59.3
  12 months; n=46 | 54.3

6. Secondary Outcome: Assisted Primary Patency
Description: Incidence of freedom from assisted primary patency at 30 days, six (6) and 12 months post-procedure, defined as a re-intervention of a stenosis (patent vessel) at the treatment site to prevent reocclusion
Time Frame: Through 12 Months
Population: 65 at 30 days; 64 at 6 months; 63 at 12 months
Measure: Number; unit: % pts free from assisted primary patency
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
% pts free from assisted primary patency
  30 days; n=65 | 100
  6 months; n=64 | 85.9
  12 months; n=63 | 76.2

7. Secondary Outcome: Assisted Secondary Patency
Description: Incidence of freedom from assisted secondary patency at 30 days, six (6) and 12 months post-procedure, defined as a re-intervention of a reocclusion (non-patent vessel) at the treatment site
Time Frame: Through 12 Month
Population: 65 at 30 days; 64 at 6 months; 63 at 12 months
Measure: Number; unit: % pts free from secondary patency
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
% pts free from secondary patency
  30 days; n=65 | 100
  6 months; n=64 | 100
  12 months; n=63 | 100

8. Secondary Outcome: Patients With >50% Stenosis Measured by Duplex Ultrasound
Description: Percentage of patients with >50% stenosis at each follow-up (30 days, six months, and 12 months post-procedure).
Time Frame: Through 12 Month
Population: per protocol; 65 patients at 30 days; 59 at 6 months and 46 at 12 months
Measure: Number; unit: percent of patients
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
percent of patients
  30 days; n=65 | 3.1
  6 months; n=59 | 40.7
  12 months; n=46 | 45.7

9. Post Hoc Outcome: Walking Impairment Questionare (WIQ)
Description: Measures difficulty in walking before and after treatment. Defined by comparing the responses to a WIQ at pre-treatment with the responses at 30 days, six (6) months and 12 months post-procedure. Higher score is better (scale 0-100).
Time Frame: measured at each follow-up period
Population: 65 patients at baseline and 30 days; 64 at 6 mo; 63 at 12 mo
Measure: Mean (Standard Deviation); unit: units on a scale 0-100
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
units on a scale 0-100
  baseline; n=65 | 45.6 (21.3)
  30 days; n=65 | 69.9 (23.7)
  6 months; n=64 | 64.7 (27.1)
  12 months; n=63 | 65.1 (25.3)

10. Secondary Outcome: Rutherford Classification
Description: Rutherford Classification at 30 days, six (6) and 12 months post-procedure. Physician assessed based on ankle pressures and treadmill testing. Rutherford scale: 0=best, 6=worst
Time Frame: Through 12 Months
Population: 63 at baseline; 62 at 30days and 6 months; 63 at 12 months
Measure: Mean (Standard Deviation); unit: units on a scale of 0-6
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
units on a scale of 0-6
  baseline; n=63 | 2.4 (0.6)
  30 days; n=62 | 1.0 (0.8)
  6 months; n=62 | 1.3 (1.1)
  12 months; n=63 | 1.3 (0.9)

11. Secondary Outcome: Adverse Events
Description: Adverse events during procedure and prior to release from the hospital, at 30 days, six (6) months, and 12 months post-procedure.
Time Frame: Through 12 Months
Measure: Number; unit: events
Arm/Group | Laser Treatment
Number analyzed (Participants) | 65
events
  Procedure/24 hours | 10
  30 days | 7
  6 months | 15
  12 months | 15
  Other | 31

12. Secondary Outcome: Volumetric Plaque Reduction
Description: Volumetric plaque reduction immediately after treatment with the CLiRpath® Photoablation Atherectomy System as determined by IVUS. Actual volume of plaque present is presented for each measurement point.
Time Frame: measured at time of procedure
Population: Per protocol
Measure: Mean (Standard Deviation); unit: millimeters cubed
Arm/Group | Laser Treatment
Number analyzed (Participants) | 48
millimeters cubed
  Post pilot channel plaque volume | 200.8 (61.0)
  Post Turbo Booster plaque volume | 192.8 (61.2)

ADVERSE EVENTS:
Arm/Group | Laser Treatment
Serious Adverse Events (participants affected / at risk) | 11/65
Other Adverse Events (participants affected / at risk) | 8/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=65)
Worsening coronary artery disease (Cardiac disorders) | 1
Right renal artery and non-treated leg stenosis (Vascular disorders) | 1
Coronary artery bypass graft (Cardiac disorders) | 2
Congestive heart failure (Cardiac disorders) | 2
Vessel occlusion (Vascular disorders) | 1
Lung cancer (Respiratory, thoracic and mediastinal disorders) | 1
Neck, back and shoulder pain (General disorders) | 1
Sternum infection (Infections and infestations) | 1
Cerebrovascular accident (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Laser Treatment (N=65)
Hematoma at access site (Surgical and medical procedures) | 4
Occlusion to treated leg other than at lesion site (Vascular disorders) | 4

LIMITATIONS AND CAVEATS:
Non-randomized study

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No